CLINICAL TRIAL: NCT05414825
Title: Monocentric Descriptive Study Regarding the Impact of Severe Dysmenorrhea on Teenagers, Their Parents and Caregivers Receiving Those Patients
Brief Title: Dysmenorrhea Exploration in Teenagers, Their Parents and Caregivers
Acronym: DEMETER
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0120
Record Dates: First submitted 2022-04-25; First posted 2022-06-10 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Dysmenorrhea
Keywords: Endometriosis; severe dysmenorrhea; pain; teenagers; pediatric; qualitative research; focus group; patient care management
MeSH Terms: conditions — Dysmenorrhea; Endometriosis; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 11 to 14 years old teenagers: Semi-structured discussion group with only young teenagers, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on the feelings of the young teenagers suffering from severe dysmenorrhea.
  Interventions: Other: focus group interview
- 15 to 17 years old teenagers: Semi-structured discussion group with older teenagers, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on the feelings of these patients suffering from severe dysmenorrhea.
  Interventions: Other: focus group interview
- 11 to 14 years old teenagers' parents: Semi-structured discussion group with parents of young teenagers, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on the feelings of the parents on the care and feelings of their child suffering from severe dysmenorrhea.
  Interventions: Other: focus group interview
- 15 to 17 years old teenagers' parents: Semi-structured discussion group with parents of older teenagers, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on the feelings of the parents on the care and feelings of their child suffering from severe dysmenorrhea.
  Interventions: Other: focus group interview
- caregivers: Semi-structured discussion group with medical staff in services potentially treating dysmenorrhea patients, moderated by a neutral facilitator in the presence of an observer, which aims to collect information on the feelings of the caregivers on the care and feelings of the patients suffering from severe dysmenorrhea.
  Interventions: Other: focus group interview

INTERVENTIONS:
Other: focus group interview — Group interview gathering words, views, symptoms and its repercussions, and main issues of the subjects regarding severe dysmenorrhea

SUMMARY:
Teenagers experimenting severe dysmenorrhea also face age-specific challenges, particularly impacting their self-confidence, self-esteem, and relations. On one hand, the study team will conduct focus group interviews to better understand the experience of teenagers and their parents consulting pediatric services for severe dysmenorrhea. On the other hand, they will conduct focus group interviews with caregivers from services that usually encounter such patients (gastrologic, gynecologic and pain services). This, allowing to later propose specific tools and healthcare organization to evaluate and accompany teenagers suffering from severe dysmenorrhea.

DETAILED DESCRIPTION:
Endometriosis is a complex disease that remains underdiagnosed (7 to 9 years delay), and incorrectly treated. While endometriosis was at first considered as a condition affecting adult women, since the early 2000s, literature has described more and more cases of adolescent patients, with frequently atypical presentations. Indirect prevalence estimates ranging from 25% to 100% in adolescents' girls with pelvic pain. Moreover, Arruda et al. indicate that adolescents girls arrive after a delay in diagnosis which has a significant impact on the progression of the disease and on their confidence in the medical listening and understanding abilities. However, the pain induced by dysmenorrhea has a profound impact on everyday life of and are frequently responsible for school missing as shown in the RESENDO survey.

By conducting a qualitative analysis based on focus groups, the main objective of the study is to describe as faithfully and extensively as possible the experience of teenage patients and their parents consulting for severe dysmenorrhea, and delineate factors potentially improving or hindering care engagement.

The study utilizes a qualitative method as a tool to have a better understanding of this population, a population increasing in pediatric gynecology services or pain management consultations. Gathering their words, their views on their symptoms and its repercussions, and their main issues, will enable to build a relationship of trust with caregivers, better address the broad problematic, and identify risk factors.

ELIGIBILITY:
INCLUSION CRITERIA :

* For " teenage" groups:

  * adolescents between 11 and 17 years old
  * consulting for severe dysmenorrhea (whether through pediatric gynecology, pain management or gastric consultation)
* For "parents" groups:

  o Parent (mother or father) of an adolescent patient consulting for severe dysmenorrhea
* For "medical staff" groups:

  * Member of a consultation receiving adolescent patients with severe dysmenorrhea
  * All type of professionals (nurses, psychologist, doctors…)

Exclusion criteria :

* For " teenage" groups:

  * suffering from an identified chronical disease
  * identified psychiatric condition
* For "parents" groups:

  o Parents whose adolescent opposes their participation in this study
* For "medical staff" groups:

  * no exclusion criteria

Ages: 11 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 3 types of population with a link to severe dysmenorrhea (whether through their own story, or child, or profession described throught eligibility criteria above)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
main themes emerging from focus group | up to one year
  qualitative outcome : identifying the main verbatim used during the focus group

CONTACTS AND LOCATIONS:
Overall Officials: Agnès SUC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Uh Toulouse, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No